CLINICAL TRIAL: NCT00608803
Title: A Phase I Study of ZIO-201-T in Combination With Doxorubicin in Subjects With Advanced, Refractory Solid Tumors for Which no Standard Therapy Exists and for Whom Treatment With Doxorubicin is Considered Medically Acceptable
Brief Title: Phase 1 Study of ZIO-201-T in Combination With Doxorubicin in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Jon Lewis, Chief Medical Officer, ZIOPHARM Oncology, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM1002
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Once the maximum tolerated dose (MTD) is determined, an expanded cohort of 20 subjects with advanced, ifosfamide and doxorubicin naive soft-tissue sarcoma subjects will be dosed at the MTD and evaluated for efficacy.
  Interventions: Drug: ZIO-201-T and doxorubicin

INTERVENTIONS:
Drug: ZIO-201-T and doxorubicin — ZIO-201-T given for 3 consecutive days every 3 weeks. Doxorubicin is given once every 3 weeks. This is a dose escalation arm.

SUMMARY:
The study of safety of ZIO-201-T in combination with doxorubicin in the treatment of advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histological or cytological documentation of cancer
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Ifosfamide and doxorubicin naïve
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements conducted within 7 days prior to dosing:Hemoglobin >9.0 g/dL, Absolute neutrophil count (ANC) >1,500/mm3,Platelet count ≥100,000/mm3,Total bilirubin <1.5×ULN,ALT and AST ≤2.5×ULN,Partial thromboplastin [PT]-INR/activated partial thromboplastin time [PTT] <1.5×ULN. Subjects who are being therapeutically anticoagulated with an agent such as Coumadin (warfarin sodium) or heparin are allowed provided there is no prior evidence of underlying abnormality in coagulation parameters. If an interaction between study drug and anticoagulant is suspected, anticoagulation monitoring should be increased as appropriate. Serum creatinine ≤ULN
* Written, informed consent must be obtained from a potential subject prior to the conduct of any study-specific procedures
* Male and female subjects must agree to use adequate birth control measures/barrier control during the course of the trial.
* Women of childbearing potential must have a pregnancy test performed within 7 days of the start of treatment.

Exclusion Criteria:

* Clinically evident congestive heart failure >Class II of the New York Heart Association (NYHA) guidelines
* Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia, or ventricular arrhythmias classified as Lown III, IV, or V
* History and/or signs of active coronary artery disease/ischemia with or without angina pectoris
* Serious myocardial dysfunction defined as scintigraphically (MUGA, myocardial scintigram) determined absolute left ventricular ejection fraction (LVEF) below 45% or an LVEF below the normal limit (one or both criteria is sufficient for exclusion)
* History of HIV infection
* Prior nephrectomy of history of urinary tract obstruction
* Active, clinically serious infection requiring systemic antibacterial, antifungal, or antiviral therapy
* Any major surgery within 3 weeks prior to start of treatment
* Metastatic brain or meningeal tumors, unless the subject is >6 months from definitive therapy and has a negative imaging study within 4 weeks of study entry. In addition, the subject must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable, provided the dose is stable for 1 month prior to study start, and following screening radiographic studies).
* History of seizure disorder (a subject with seizures related to brain metastasis will be allowed provided he/she has been seizure-free for at least 2 months and meets the criteria defined above for inclusion of subjects with brain metastasis)
* Previous malignancy (except cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis, & T1] or other malignancies curatively treated >3 years prior to entry)
* Pregnancy or lactation
* Substance abuse or medical, psychological, or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Any condition that is unstable or could jeopardize the safety of a subject and his/her compliance with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Toxicities | 5 months

SECONDARY OUTCOMES:
Pharmacokinetics | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, Study Director — ZIOPHARM Oncology, Inc.
Locations (2):
- United States (2):
  - Santa Monica, California
  - Houston, Texas